CLINICAL TRIAL: NCT02708459
Title: Transversus Abdominus Plane Block in Living Donor Hepatectomy
Acronym: TAP Donor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AlRefaey Kandeel (Other)
Responsible Party: Sponsor-Investigator, AlRefaey Kandeel, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Abuelella TAP
Record Dates: First submitted 2016-02-09; First posted 2016-03-15 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Living Donor Hepatectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): Control group where postoperative analgesia will be maintained by Morphine intravenous boluses (2 mg) if Visual analogue scale (VAS) scale more than 4.
  Interventions: Drug: Intravenous morphine
- Bupevecaine group (Active Comparator): Postoperative analgesia will be maintained by 20 ml Bupevecaine (0.25%) boluses in surgically inserted TAP catheter each 8 hours for 48 hours with rescue analgesia intravenous morphine (2mg) if VAS more than 4
  Interventions: Device: surgically inserted Transversus abdominus plane catheter; Drug: Intravenous morphine; Drug: Bupevecaine
- Dex group (Active Comparator): catheter will surgically inserted in Transversus abdominus plane (TAP) plane before wound closure Postoperative analgesia will be maintained by Dexmedetomedine 0.4 mg/kg plus Bupevecaine 0.25 20 ml boluses each 8 hours for 48 hours in surgically inserted TAP catheter with rescue analgesia intravenous morphine (2mg) if VAS more 4
  Interventions: Device: surgically inserted Transversus abdominus plane catheter; Drug: Intravenous morphine; Drug: Bupevecaine; Drug: Dexmedetomedine

INTERVENTIONS:
Device: surgically inserted Transversus abdominus plane catheter — at end of surgery, a surgeon will insert catheter in Transversus abdominus plane (TAP) between internal oblique muscle and Transversus abdominus muscle
  Arms: Bupevecaine group; Dex group
Drug: Intravenous morphine — Boluses of intravenous morphine (2 mg) will be given to patients if Visual analogue scale (VAS) more than 3
Drug: Bupevecaine
  Arms: Bupevecaine group; Dex group
Drug: Dexmedetomedine
  Arms: Dex group

SUMMARY:
Comparing different drugs used in Transversus abdominus plane analgesia after donor hepatectomy. Patients will be divided into three groups; control group, Bupivecaine group, and Dexmedetomedine group according to the used drug

DETAILED DESCRIPTION:
Transversus abdominus plane block for postoperative analgesia after donor hpatectomy surgery using three different drugs control group, Bupivecaine group, and Dexmedetomedine group

ELIGIBILITY:
Inclusion Criteria:

* all living hepatectomy donors in Mansoura liver transplantation program

Exclusion Criteria:

* refusal known sensetivity to used drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
postoperative morphine (mg) consumption in 1st 48 hours | 48 hours postoperative

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura university, Al Mansurah, Dakahlia Governorate
  - Mansoura university, Al Mansurah, Dkahleya

IPD SHARING:
Plan to Share IPD: Yes